CLINICAL TRIAL: NCT03057704
Title: Comparison of Two Techniques of Administering IV Lidocaine in Reducing Propofol Injection Pain
Brief Title: Comparison of Two Techniques of IV Lidocaine on Propofol Injection Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00040756
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Results first posted 2018-02-13 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Injections, Intravenous
Keywords: Propofol; lidocaine; pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Tourniquets

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial of two methods of administering lidocaine prior to propofol injection
Who Masked: Participant
Masking Description: The participant is not told which group they are randomized to. However, a tourniquet is applied in the experimental group, thus some subjects may reason that they are in the experimental group. The study coordinator is aware which group the subject is in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intravenous lidocaine: flushed (Active Comparator): Lidocaine injection flushed
  Interventions: Drug: Lidocaine injection flushed
- Intravenous lidocaine: tourniquet (Experimental): Lidocaine injection tourniquet
  Interventions: Drug: Lidocaine injection tourniquet

INTERVENTIONS:
Drug: Lidocaine injection flushed — The investigator administers IV lidocaine and flushes it into the subject prior to administering propofol.
  Other Names: Xylocaine
  Arms: Intravenous lidocaine: flushed
Drug: Lidocaine injection tourniquet — Intravenous lidocaine: tourniquet
  Other Names: Xylocaine; Tourniquet
  Arms: Intravenous lidocaine: tourniquet

SUMMARY:
Intravenous lidocaine is commonly given through an intravenous (IV) line prior to injection of propofol to reduce the amount of pain during propofol injection. The investigators want to study if giving the lidocaine through the IV while the forearm on the same limb has a tourniquet applied to it to prevent "washing out" of the lidocaine prior to propofol injection helps reduce propofol injection pain.

DETAILED DESCRIPTION:
The investigators expect that tourniquet lidocaine is superior to straight non-tourniquet lidocaine in reducing propofol injection pain. The investigators also wanted to determine the association of tourniquet duration on reduction of pain with propofol administration. Small studies indicate that 60 seconds of tourniquet lidocaine is superior to 30 seconds or less of tourniquet duration or mixed lidocaine/propofol for injection. The investigators suspect many clinicians do not use the 60-second tourniquet technique due to the extra time involved but hypothesize that a more practical application by applying the tourniquet as soon as the patient is positioned on the operating table will not only be more widely adopted by clinicians as it does not cause delay but also provide the necessary amount of time for benefit from the tourniquet. The investigators also wanted to record the time from tourniquet application to start of propofol administration, which the investigators predict would be at least 60 seconds to see if there is a correlation between duration of venous stasis of IV lidocaine and pain benefit.

Methods and Measures

Design This was conducted as a randomized controlled trial of two methods of administering lidocaine prior to propofol injection.

Setting The study setting was located within North Carolina Baptist Health, an academic medical center, in the Endoscopy Suite or Outpatient Surgery Center where subjects were scheduled to receive propofol as part of their sedation or anesthetic.

Sample Size The investigators estimated that 25 subjects in each of the two groups was required to test the hypothesis based on prior studies.

Interventions and Interactions

The investigators used two groups:

* Group 1: 50mg of 2% lidocaine given just prior to the propofol dose through the IV line.
* Group 2: 50mg of 2% lidocaine given IV with venous occlusion applied when the patient is positioned on the operating room table and timed until the onset of propofol administration. The tourniquet the investigators used was a Quick Release tourniquet applied to the forearm 10cm distal to the elbow joint in the tourniquet group. Venous stasis was confirmed with cessation of flow from hanging IV fluid.

For both groups, no premedication was given, which is the normal practice for these procedures. Study procedures involved placing a 20 gauge intravenous (IV) catheter in a vein distal to the mid forearm. Venous occlusion was achieved by either a latex free tourniquet or McKesson Quick Release tourniquet applied to the forearm 10cm distal to the elbow joint. Tourniquet pressure was somewhat variable but sufficient to cause venous stasis as confirmed by no flow of hanging IV fluid. Injections were delivered at roughly 1 ml/sec.

Schedule of events in the study (all performed by 1 of the 2 investigators:

* Day of procedure: holding area

  * Consent subject for study participation
  * Randomly assign patient to one of two groups
* Day of procedure: procedure area

  -Accompany subject to the operating or procedure room, perform protocol from the group to which the subjects were assigned, while noting outcome measures such as self-described discomfort and observer graded discomfort
* Day of procedure: recovery area

  -Revisit subject in recovery 30 minutes after their procedure to determine post-procedure recall of discomfort
* Post-study period
* Analyze data

Analytical Plan The investigators will analyze results initially using descriptive statistics. Comparison between groups was done using chi square tests for proportions, and t-tests or ANOVA procedures for continuous variables. Regression analysis was performed to identify independent outcome predictors. Other inferential statistical analysis was conducted as appropriate.

Informed Consent One of the two investigators obtained signed informed consent from each subject. This was performed in the holding room prior to the procedure since most subjects had their pre-procedure examination performed in the holding room and were not seen prior to the day of their procedure.

ELIGIBILITY:
Inclusion Criteria:

* Any subject at North Carolina Baptist Hospital scheduled for a procedure in which they will receive propofol for sedation or anesthesia and will not be receiving any other medications prior to the propofol injection.
* Cases must be schedule to have a duration less than 60 minutes.

Exclusion Criteria:

* Subjects are excluded if they cannot verbalize a rating of pain
* Subjects are excluded if they require intravenous medications prior to the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy N Harwood, MD, Principal Investigator — Wake Forest University Health Sciences; Patrick Grace, MD, Study Director — Wake Forest University Health Sciences
Locations (1):
- North Carolina Baptist Hospital, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were approached after they were scheduled for colonoscopy or minor procedures and appeared in the holding area for procedures in which propofol sedation or induction of general anesthesia was used.
Period: Overall Study
Arm/Group | Intravenous Lidocaine: Flushed | Intravenous Lidocaine: Tourniquet
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects were eligible is schedule for procedures in which they would receive propofol for sedation or induction. Subjects included a general local population from the Piedmont Triad of North Carolina.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Lidocaine: Flushed | Intravenous Lidocaine: Tourniquet | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (6.9) | 54 (7.3) | 53 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Pain score at IV prior to procedure [Count of Participants; unit: Participants]
  IV pain score of 0 | 25 | 25 | 50
  IV pain score of 1-3 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Expression of Pain
Description: Patient's verbal rating of pain during injection (see link to study protocol)
  We used a Verbal Rating Scale from the patient that self-described discomfort level during injection using question:
  How would you rate your pain using None, Mild, Moderate, Severe and record it on this 4-point scale:
  * None (0)
  * Mild (1)
  * Moderate (2)
  * Severe (3) None is no pain (best outcome) and Severe is worst pain possible (worst outcome).
Time Frame: During injection at beginning of study; lasts 10 seconds one time only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Lidocaine: Flushed | Intravenous Lidocaine: Tourniquet
Number analyzed (Participants) | 25 | 25
units on a scale | 0.76 (1.0) | 0.04 (0.2)

2. Secondary Outcome: Subject's Recall of Injection Discomfort
Description: Investigator asks patient if they recall discomfort during injection after the procedure.
  Patient's verbal rating and recall of pain during injection.
  We used a Verbal Rating Scale from the patient that self-described discomfort level during injection using question:
  How would you rate your pain using None, Mild, Moderate, Severe and record it on this 4-point scale:
  * None (0)
  * Mild (1)
  * Moderate (2)
  * Severe (3) None is no pain (best outcome) and Severe is worst pain possible (worst outcome).
Time Frame: This occurs 30 minutes after the subject's procedure is finished in the recovery room; lasts 30 seconds one time only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Lidocaine: Flushed | Intravenous Lidocaine: Tourniquet
Number analyzed (Participants) | 25 | 25
units on a scale | 0.52 (0.82) | 0.04 (0.2)

3. Secondary Outcome: Investigators Rating of Patient Discomfort
Description: Investigator rates patient's nonverbal display of discomfort.
  Investigator Assessments:
  Induction Discomfort Scale (during injection and within 5 seconds after injection)
  * No change in patient behavior (0)
  * Grimace (1)
  * IV forearm withdrawal (2)
  * Moaning (3)
  * Verbal statement of discomfort ("it hurts", etc.) (4) 0 indicates desired outcome of no pain and 4 indicates worst IV pain experienced.
Time Frame: During injection at beginning of study period; lasts 10 seconds one time only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Lidocaine: Flushed | Intravenous Lidocaine: Tourniquet
Number analyzed (Participants) | 25 | 25
units on a scale | 1.12 (1.27) | 0 (0)

ADVERSE EVENTS:
Time Frame: We studied the subjects in this time frame: 1) Initiated contact with them in the holding area just prior to their procedure. 2) We assessed their verbal expression of discomfort and their display of discomfort (outcomes 1 and 2) during propofol injection and up to 30 seconds after injection 3) We assessed their recall of discomfort approximately 30 minutes after their procedure while they were in the recovery area. 4) They were then discharged home without further involvement in the trial.
Description: Patients were interviewed in the recovery room at least 30 minutes after their procedure by one of the investigators, and they were called the next business day by a recovery room nurse for followup and asked about any adverse events they experienced after discharge.
Arm/Group | Intravenous Lidocaine: Flushed | Intravenous Lidocaine: Tourniquet
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Results became clear at total number of subject =25.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03057704/Prot_SAP_ICF_000.pdf